CLINICAL TRIAL: NCT07157020
Title: A Multi-center and Multidisciplinary Research Project on Prevention, Early Detection, and Clinical Evaluation of Intracranial Hemorrhage in Preterm Infants
Brief Title: Research on Prevention, Early Detection, and Clinical Evaluation of Intracranial Hemorrhage in Preterm Infants
Acronym: ROPEDACEOIHIPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2025-06-108
Record Dates: First submitted 2025-08-26; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Intraventricular Hemorrhage of Prematurity
Keywords: Intraventricular Hemorrhage of Prematurity; prevention; early detection; clinical evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-threshold intervention group (Experimental): VI>P97，but ≤ P97+4mm
  Interventions: Procedure: ommaya capsule implantation technique
- high-threshold intervention group (Experimental): VI>P97+4mm
  Interventions: Procedure: ommaya capsule implantation technique

INTERVENTIONS:
Procedure: ommaya capsule implantation technique — Intervention criteria: Low-threshold intervention group and high--threshold intervention group
  Other Names: Lumbar puncture drainage

SUMMARY:
1. Establish a reference curve for the lateral ventricular diameter of premature infants and determine the intervention threshold for hydrocephalus after hemorrhage in premature infants based on the reference curve, providing a scientific basis for optimizing clinical intervention.
2. Apply ultrasound radiomics technology to explore and formulate new standards for imaging diagnosis and treatment; By integrating metabolomics, ultrasound radiomics and clinical data, high-risk individuals for intracranial hemorrhage and their relationship with prognosis can be identified early.
3. To explore whether advancing the indication for surgical intervention of hydrocephalus in preterm infants after hemorrhage from ventricular index P97+4mm to P97 and whether repeated lumbar puncture and drainage can improve their prognosis, with the aim of clarifying the optimal timing for intervention of hydrocephalus in preterm infants after hemorrhage and optimizing the treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 23+0 weeks to 36+6 weeks;
* Post-hemorrhagic hydrocephalus is confirmed by cranial ultrasound or other cranial imaging examinations.
* No cerebrospinal fluid drainage treatment was received before enrollment.

Exclusion Criteria:

* Excluding secondary IVH, including but not limited to congenital malformations, vitamin K1 deficiency, abnormal coagulation function, etc.
* Excluding hydrocephalus caused by other reasons, including but not limited to infection, congenital malformations, intracranial space-occupying lesions, etc.
* Treatment before diagnosis of hydrocephalus after intraventricular hemorrhage or suspected presence of central nervous system infection.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Death or the occurrence of neurodevelopmental disorders (NDI) before the corrected gestational age of 2 years. | The assessment times are CA at 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months respectively.
  NDI can be diagnosed if any of the following conditions are met.
  * Cerebral palsy;
    * Griffiths score <85 points for the corresponding age: The assessment times are CA at 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months respectively. Any assessment score lower than 85 points is considered a positive event.
      * Sensorineural or mixed hearing impairment and non-congenital hearing loss require hearing AIDS or cochlear implants
        ④ Bilateral visual impairment;
        * Epilepsy.

IPD SHARING:
Plan to Share IPD: No